CLINICAL TRIAL: NCT01789853
Title: Improving the Delivery of Intensive Gait Training in the Clinical Setting to Augment Community Ambulation
Brief Title: Very Intensive Early Walking in Stroke
Acronym: VIEWS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shirley Ryan AbilityLab (Other)
Responsible Party: Principal Investigator, T. George Hornby, T. George Hornby, PT, PhD, Shirley Ryan AbilityLab
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STU00010421
Record Dates: First submitted 2012-05-14; First posted 2013-02-12 (Estimated); Last update posted 2015-09-09 (Estimated); Status verified 2015-09

CONDITIONS: Stroke
Keywords: stroke, rehabilitation, gait training
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intensive Walking (Experimental): High intensity walking training in variable context for 8 weeks
  Interventions: Behavioral: Intensive Walking
- Conventional Physical Therapy (Active Comparator): Regular physical therapy for 8 weeks
  Interventions: Behavioral: Conventional Physical Therapy

INTERVENTIONS:
Behavioral: Intensive Walking — 8 weeks high intensity walking training over multiple stepping tasks
  Arms: Intensive Walking
Behavioral: Conventional Physical Therapy — Regular physical therapy for 8 weeks
  Arms: Conventional Physical Therapy

SUMMARY:
The purpose of this study is to demonstrate the efficacy of intensive locomotor interventions early post stroke. An intensive locomotor training (LT) program will be compared to an active control, conventional physical therapy. It is proposed that an early and intensive stepping paradigm that is not typically employed early in physical therapy will lead to superior outcomes and improved community mobility. A randomized, blinded, controlled trial will test subjects with moderate to severe locomotor dysfunction in individuals post-stroke to compare walking-related outcomes after intensive gait training (including treadmill, overground, stair training, and skilled walking training) to outcomes after conventional physical therapy.

DETAILED DESCRIPTION:
In Aim 2, intensive gait training overground and on the treadmill using the device as appropriate will be provided using a randomized, controlled trial (RCT) design. Determination of optimal swing phase and propulsive assistance provided to subjects to maximize treadmill walking velocity (in Aim 1) will be necessary to assess the efficacy of this technique to improve walking function over prolonged LT sessions. Consistent with work from the previous grant cycle12, we will compare the relative improvements in impairments, activity and participation following 1 of 2, 8 -week interventions to improve walking ability post-stroke. Fifty-six (56) subjects will be recruited, stratified based on walking 10 meters [requiring moderate assistance (subject performing 50-74%), minimal assistance (subject performing greater than 75% of gait but still needing assist), with a gait speed <0.5m/s without assist, or with gait speed of >0.5-0.9m/s without assist. Subjects will be randomized to experimental (intensive gait training using aforementioned gait training principles) or control conditions (conventional physical therapy). The test group will receive 40, 40-minute LT sessions during a 60 minute time period over 8 weeks with subjects ambulating on the treadmill, overground, and on stairs. During the first 5 training sessions, LT will take place solely on the treadmill. After that time, half of the sessions will be walking overground and stairs and half on the treadmill. Training will be performed with a target heart rate of 70-80% of heart rate reserve (HRR) and subjective ratings of perceived exertion of 14-17 when patients are on medications to limit heart rate kinetics. Kinematics during LT will be monitored visually to ensure proper foot placement necessary for continuous stepping while maintaining the appropriate intensity, using the device as necessary. The control group will receive conventional physical therapy (receiving at least 3 sessions of physical therapy per week) at the subject's and medical teams' discretion (day rehabilitation, outpatient, or home health). If the subject is not receiving at least 3 sessions of physical therapy per week, control therapy treatments will be provided consistent with recent data detailing the amount of specific physical therapy activities provided during single-session outpatient visits19and published data21 as well as unpublished data from Moore that delineates the number of steps taken per conventional therapy session based on the gait speed of individual (number of steps during training=1500*gait speed+200). The additional 200 steps were added to this algorithm to allow for individuals who require assist to receive gait training during the sessions. Clinical and quantitative assessment of neuromuscular and cardiopulmonary impairments, limitations in activity and participation, assessment of corticospinal tract (CST) excitability and integrity will be performed prior to training, mid-training, end of 8 week training, and with a 2-6 month follow-up examination. Control group participants will have the option of participating in 4 weeks of intensive gait training (experimental protocol) at the end of the follow up testing and complete one more testing session at the end of those 4 weeks. Primary outcome measures include laboratory and community measures of ambulatory function, including gait speed over short distances, distance walked and gait efficiency during the 6 min walk, and the amount of daily community stepping (using Step Activity Monitors [SAM]20), CST excitability measures using transcranial magnetic stimulation (TMS) (optional) and assessment of white matter tract integrity using MRI (optional).

ELIGIBILITY:
Inclusion Criteria:

* subacute (<6 months) stroke
* 18-75 years old
* history of history of unilateral, supratentorial, ischemic or hemorrhage stroke
* able to walk 10m without physical assistance
* gait speed less than or equal to .8m/s
* medical clearance

Exclusion Criteria:

* significant cardiorespiratory or metabolic disease that may limit exercise participation
* weight limit > 250 lbs (limit of most counter-weight safety systems)
* history of previous orthopedic or neurological conditions which may impair walking.
* women of childbearing potential will not be excluded, although women who are pregnant will be excluded due to potential forces at trunk from the harness applied at the waist.
* subjects with scores < 23 on the Mini Mental Status Exam

  * Exclusion for transcranial magnetic stimulation (TMS):
* pacemaker
* metal implants in the head region
* history of epilepsy or seizures
* skull fractures or skull deficits
* concussion within the last 6 months
* unexplained recurring headaches
* medications that lower seizure threshold
* pregnancy

  * Exclusion for the MRI:
* aneurysm clip or coil
* metal or wire implants
* heart valve prosthesis

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2008-10; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Change in 10 meter walk test | Pre Test, 4 weeks, 8 weeks, 3 month follow up
  Gait speed

SECONDARY OUTCOMES:
Change in 6 min walk test | 0, 4, 8 weeks post-training and 2 month follow-up
  Timed walking distance over 6 min at self-selected speed
Change in Berg Balance Scale | 0. 4. 8 weeks post-training and 2 month follow-up
  Standardized balance assessment

CONTACTS AND LOCATIONS:
Overall Officials: George T Hornby, PT, PhD, Principal Investigator — Shirley Ryan AbilityLab
Locations (1):
- Rehabilitation Institute of Chicago, Chicago, Illinois, United States

REFERENCES:
- [Derived] Hornby TG, Rafferty MR, Pinto D, French D, Jordan N. Cost-Effectiveness of High-intensity Training vs Conventional Therapy for Individuals With Subacute Stroke. Arch Phys Med Rehabil. 2022 Jul;103(7S):S197-S204. doi: 10.1016/j.apmr.2021.05.017. Epub 2021 Jul 3. PMID 34228956
- [Derived] Hornby TG, Henderson CE, Holleran CL, Lovell L, Roth EJ, Jang JH. Stepwise Regression and Latent Profile Analyses of Locomotor Outcomes Poststroke. Stroke. 2020 Oct;51(10):3074-3082. doi: 10.1161/STROKEAHA.120.031065. Epub 2020 Sep 4. PMID 32883192
- [Derived] Hornby TG, Holleran CL, Hennessy PW, Leddy AL, Connolly M, Camardo J, Woodward J, Mahtani G, Lovell L, Roth EJ. Variable Intensive Early Walking Poststroke (VIEWS): A Randomized Controlled Trial. Neurorehabil Neural Repair. 2016 Jun;30(5):440-50. doi: 10.1177/1545968315604396. Epub 2015 Sep 3. PMID 26338433